CLINICAL TRIAL: NCT01436916
Title: Oral Cholecalciferol in Prevention of Type 2 DM in Prediabetic Population With Vitamin D Insufficiency
Brief Title: Oral Cholecalciferol in Prevention of Type 2 Diabetes Mellitus
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Post Graduate Institute of Medical Education and Research, Chandigarh (Other)
Responsible Party: Principal Investigator, Anil Bhansali, professor and head of the department of Endocrinology, Post Graduate Institute of Medical Education and Research, Chandigarh
Organization: PIMERIndia (Unknown)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 0023051981
Record Dates: First submitted 2011-09-13; First posted 2011-09-20 (Estimated); Last update posted 2015-10-26 (Estimated); Status verified 2015-10

CONDITIONS: Prediabetes; Vitamin D Deficiency
Keywords: prediabetes; oral cholecalciferol
MeSH Terms: conditions — Prediabetic State; Vitamin D Deficiency | interventions — Cholecalciferol

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- oral cholecalciferol + lifestyle counselling (Active Comparator): will receive Oral cholecalciferol
  Interventions: Drug: oral cholecalciferol + life style counselling
- Placebo + lifestyle counselling (Placebo Comparator): will receive placebo
  Interventions: Drug: placebo + life style counselling

INTERVENTIONS:
Drug: oral cholecalciferol + life style counselling — oral cholecalciferol 600000 units loading then 60000 units fortnightly for 6months
  Arms: oral cholecalciferol + lifestyle counselling
Drug: placebo + life style counselling — Will provide placebo 10 sachets loading and then single sachet fortnightly for 6 months
  Arms: Placebo + lifestyle counselling

SUMMARY:
Type 2 diabetes mellitus (T2DM) is a major public health problem .Prevalence of vitamin D deficiency is also high i.e. 78-96% in different groups of population in north India. Observational studies find association between low Vitamin D status and type 2 diabetes mellitus. Prediabetes is a condition that progress to diabetes at a rate of 6-10% per year .There is mechanistic support that vitamin D may influence both insulin secretion and insulin sensitivity and subsequently T2DM incidence. In general, cross-sectional and prospective studies support the role of vitamin D in the prevention of T2DM. This study will be a single blind randomized placebo controlled trial to study the effect of oral cholecalciferol in insulin sensitivity and secretion in adults with prediabetes who are also vitamin D insufficient.

ELIGIBILITY:
Inclusion Criteria:

* Adults > 20 years
* Impaired fasting glucose (IFG) - FPG 100-125 mg/dl
* Impaired glucose tolerance((IGT)- 2hr PPG 140-199mg/dl

OR

* both ( IFG +IGT)
* with or without Hb A1c -5.7-6.4 %

WITH

* Asymptomatic Vitamin D deficiency(< 20ng/ml) or vitamin D in sufficiency(< 32ng/ml)

Exclusion Criteria:

* Diabetes mellitus,
* Base line 25(OH)D3 > 32 ng/ml,
* Symptomatic vitamin D deficiency,
* Any medication within last month that could affect insulin secretion, insulin sensitivity , vitamin D and calcium metabolism
* Chronic renal , hepatic ,malignant, intestinal or endocrine diseases
* Febrile illness or infective morbidity in last 2 weeks,
* Grossly deranged liver and kidney function

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2011-09; Primary Completion 2012-09 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Change in insulin sensitivity using OGIS (oral glucose insulin sensitivity index) | Base line and 6 months

SECONDARY OUTCOMES:
change in indices of insulin secretion using HOMA1-beta% and HOMA2-beta % | Base line and 6 months
change in other insulin sensitivity indices | Base line and 6 months
  QUICKI, HOMA 1-IR ,HOMA2- IR ,WBISI( Matsuda index),hepatic and muscle insulin sensitvity indices
Change in Hb A1c | Base line and 6 months
Change in fasting and post prandial blood glucose | 0,3, 6months

CONTACTS AND LOCATIONS:
Overall Officials: Anil Bhansali, MD, DM, Principal Investigator — Post Graduate Institute of Medical Education and Research, Chandigarh
Locations (1):
- PGIMER, Chandigarh, Chandigarh(UT), India